CLINICAL TRIAL: NCT00411307
Title: A Randomized, Open-Label, Single-Dose, Pilot Study to Evaluate the Safety and Efficacy of OROS Hydromorphone in Patients With Acute, Moderate-to-Severe Postoperative Pain
Brief Title: A Randomized, Open-Label, Single-Dose, Small Study to Evaluate the Safety and Effectiveness of Hydromorphone in Patients With Short Term, Moderate to Severe Postoperative Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alza Corporation, DE, USA (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR013267
Record Dates: First submitted 2006-12-12; First posted 2006-12-14 (Estimated); Last update posted 2010-04-27 (Estimated); Status verified 2010-04

CONDITIONS: Pain, Postoperative; Orthopedic Procedures; Analgesia
Keywords: Analgesia; Postoperative pain
MeSH Terms: conditions — Pain, Postoperative; Agnosia

INTERVENTIONS:
Drug: OROS hydromorphone HCI

SUMMARY:
The purpose of this small study was to investigate the safety and effectiveness of OROS hydromorphone HCI for the treatment of short-term, moderate to severe postoperative pain following total knee replacement surgery.

DETAILED DESCRIPTION:
This was a multicenter, randomized (patients are assigned different treatments based on chance), open-label, single dose small study. During the 36 hour study period, concomitant analgesic (pain) medications and physical therapy were recorded in the patient's case report form. The study duration for each patient was 36 hours after a single dose of OROS hydromorphone HCI had been administered. After surgery, eligible patients had to tolerate liquids, swallow a tablet, and have audible bowel sounds. Before OROS hydromorphone HCI was administered, all analgesic medications were discontinued and patients with a pain score of 2(moderate pain) or 3 (severe pain) upon movement were eligible to enter the study and receive a single oral dose of OROS hydromorphone HCI. Patients had to have stable heart rates, blood pressure, respiration, oxygen saturation greater than or equal to 94% and patients who had undergone regional anesthesia had to have motor and sensory recovery from nerve blockade. Qualifying patients were given OROS hydromorphone HCI between 6 and 48 hours after completion of the surgical procedure. Patients were randomized into 3 groups (OROS hydromorphone HCI 8, 16, and 32 mg). The precise time of OROS hydromorphone HCI administration was considered time zero. To maintain consistency, dosing was to occur between 6 am and 2 pm, if possible. Following study drug administration, patients could be given rescue medication of oral hydromorphone immediate-release tablets (2 or 4 mg) for breakthrough pain as needed. Oxygen saturation, vital signs, pain relief ratings, and pain intensity ratings at rest and upon movement were obtained at 2-hour time intervals during the first 8 hours following study drug administration, and at 4 hour intervals from 8 to 36 hours following study drug administration. The study concluded 36 hours after dosing, at which time a global evaluation of pain relief was obtained from each patient. One single dose of OROS hydromorphone HCI (8, 16, or 32 mg) administered orally at the beginning of the 36 hour study.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing primary, unilateral total knee replacement surgery where use of opioid analgesics for short-term postoperative pain is required
* At baseline must be able to tolerate oral liquids, swallow a tablet, and have the presence of bowel sounds upon examination
* Patients must demonstrate stable vital signs immediately before dosing with OROS hydromorphone HCI
* At baseline pain intensity upon movement must be scored by the patient as 2 or 3 (moderate or severe) on the Pain Intensity Rating Scale
* At baseline patients receiving regional anesthetics/analgesics must demonstrate recovery from the motor and sensory effects of the nerve blockade
* Patients must be administered OROS hydromorphone HCI between 6 and 48 hours following completion of surgery
* Patients should expect to remain hospitalized for 36 hours after study drug administration.

Exclusion Criteria:

* Patients either intolerant of hydromorphone or who have experienced an anaphylactic IgE-mediated immune response (e.g. hives, wheezing, angioedema or bronchospasms) to any opioid agonist
* Patients having previously undergone the following major surgery for high tibial osteotomy, knee arthroplasty to the affected knee
* Patients with any gastrointestinal disorder, including pre-existing severe GI narrowing (pathologic or iatrogenic) that may affect the absorption or transit of orally administered drugs
* Patients who are pregnant or breast-feeding. A negative pregnancy test is required prior to administration of the study medication in females of childbearing potential
* Patients with significant CNS disorder, including but not limited to head injury, intracranial lesion, increased intracranial pressure, seizure disorder, stroke within the past 6 months, and disorders of cognition
* Patients with clinically significant impaired renal, hepatic, or hematological function
* adrenocortical insufficiency
* uncontrolled hypothyroidism or hyperthyroidism, or clinically significant urinary obstruction

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Study Completion 2001-10 (Actual)

PRIMARY OUTCOMES:
Variables measured included: Total number of doses/amount of rescue medication hydromorphone (immediate release) taken for breakthrough pain during 36 hours post OROS hydromorphone (slow release) administration

SECONDARY OUTCOMES:
Variables measured included:Pain relief scores; Pain intensity scores;Patient's rating of sleep interference;global evaluation of analgesia; oxygen saturation; vital signs and adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Alza Corporation Clinical Trial, Study Director — ALZA